CLINICAL TRIAL: NCT05744635
Title: Assessment of the Pharmacokinetic Profile of Tacrolimus Medications in Liver Transplant Patients
Brief Title: Assessment of the Pharmacokinetic Profile of Tacrolimus Medications and Their Relation to Effectiveness and Safety in Liver Transplant Patients
Acronym: LTA
Status: Recruiting | Type: Observational
Sponsor: Chiesi Hungary Ltd. (Industry)
Collaborators: Chiesi Slovenija, d.o.o. (Industry)
Responsible Party: Sponsor
Other Study IDs: LTA_2022
Record Dates: First submitted 2023-01-30; First posted 2023-02-27 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Liver Failure
Keywords: Liver transplantation; Immunosuppression; Tacrolimus
MeSH Terms: conditions — Liver Failure | interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Liver transplant patients, receiving tacrolimus containing immunosuppression: 1. Patients ≥ 18 years of age
  2. Patients after liver- or simultaneous liver and kidney transplantation
  3. Having received a tacrolimus containing immunosuppressant therapeutic regimen at least for four weeks (induction therapy), and TL is within 5-20 ng/ml before inclusion. Possible medications are the following (dosages and administration according to local (European) SmPC
     * Envarsus prolonged release tablet
     * Adport hard capsule
     * Advagraf prolonged-release hard capsule
     * Modigraf granule for oral suspension
     * Prograf hard capsule
     * Tacforius hard capsule
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus received as part of routine clinical care

SUMMARY:
The goal of this observational study is oo compare the pharmacokinetic parameters of different tacrolimus containing medications in liver transplant patients. The main question[s] it aims to answer are:

* Differences in pharmacokinetic parameters of tacrolimus containing medicinal products (TL, TDD and their ratio - C/D)
* Changes in liver function parameters compared to baseline.
* Change in the estimated glomerular filtration rate (eGFR) compared to baseline.
* To assess the possible relation of liver function parameters and eGFR to C/D (blood concentration and daily dosage)
* Incidence of acute graft rejection during the study
* Incidence of BK and cytomegalovirus (CMV) infection during the study
* To assess the intraindividual variability of the TL, TDD and the ratios of these parameters (C/D)
* To assess the patient-adherence of therapy based on the BAASIS questionnaire, and prescription filled by individual patients, based on electronic health-care record.

Participants will not have to undergo any additional clinical visits or tests except which are required in routine clinical care

DETAILED DESCRIPTION:
The primary aim of the study is to assess tolerability of LCPT and graft function within the 24-month observational period. Other objectives include the assessment of the intraindividual variability of the TL and TDD, the incidence of BK and cytomegalovirus infections, the incidence of graft insufficiency and acute and chronic graft rejection. There are few real-life studies available on maintenance treatment regimens in liver transplant patients throughout Europe, and these only focus on the healthcare resources' consumption. There is a lack of data describing the effectiveness of different drugs and their combinations in early maintenance immunosuppression in the real-life setting. Even less data is available of ISU (immunosuppression) drugs combinations' metabolism and its relation to effectiveness and safety, measured in liver transplant patients.

Given the above considerations we planned this non-interventional study (NIS) to assess pharmacokinetic parameters of LCPT and other tacrolimus containing medications and their relation to efficacy and tolerability in hepatic allograft recipients in a real-life setting.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age
2. Patients after liver- or simultaneous liver and kidney transplantation
3. Having received a tacrolimus containing immunosuppressant therapeutic regimen at least for four weeks (induction therapy), and TL is within 5-20 ng/ml before inclusion
4. Patients signed an informed consent form for use of their pseudonymised clinical data within the present non-interventional trial.

Exclusion Criteria:

1. Participation in any clinical trial, 30 days prior to inclusion
2. The patients received liver allograft more than 6 months before inclusion
3. Hospitalisation due to infection, acute rejection, or graft disfunction 2 weeks prior to enrolment
4. Chronic graft insufficiency in the patient's history
5. Use of medications 2 weeks prior to enrolment, or the need for continuous use of medications that are known to significantly affect the pharmacokinetics of tacrolimus containing medications (as CYP3A4 inducers: rifampin, carbamazepine, phenobarbital, and phenytoin, or CYP3A4 inhibitors: erythromycin, ketoconazole, clarithromycin, and verapamil containing medication)
6. Presence of the following comorbidities:

   1. Diseases affecting adherence to therapy (Chronic neurologic conditions, Psychiatric diseases)
   2. Diseases affecting drug absorption and metabolism (Inflammatory bowel disease, Chronic inflammatory diseases of bile ducts, Presence of ascites due to any disease)
7. Patients on waiting list for re-transplantation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult, liver (or concomittant liver-renal) transplant patients, receiving tacrolimus containing medications.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic profile TL | 12 months
  To compare the trough level (TL) of different tacrolimus containing medications to Envarsus at each visit
Pharmacokinetic profile TDD | 12 months
  To compare the total daily dose (TDD) of different tacrolimus containing medications to Envarsus at each visit
Pharmacokinetic profile C/D | 12 months
  To compare the ration of TL and TDD (C/D) of different tacrolimus containing medications to Envarsus at each visit

SECONDARY OUTCOMES:
Liver function GGT | 12 months
  Changes in Gamma glutamine transferase (GGT) levels compared to baseline.
Liver function AP | 12 months
  Changes in Alcalic phosphatase (AP) levels compared to baseline.
Liver function GOT | 12 months
  Changes in Glutamyl oxaloacetic transaminase (GOT) levels compared to baseline.
Liver function GPT | 12 months
  Changes in Glutamyl pyruvic transaminase (GPT) levels compared to baseline.
Renal function | 12 months
  Change in the estimated glomerular filtration rate (eGFR) compared to baseline.
Kinetics and function | 12 months
  To assess the possible relation of liver function parameters and eGFR to C/D (blood concentration and daily dosage)
Rejection | 12 months
  Incidence of acute graft rejection during the study
Virus infection | 12 months
  Incidence of BK and cytomegalovirus (CMV) infection during the study
Variability | 12 months
  To assess the intraindividual variability of the TL, TDD and the ratios of these parameters (C/D)
Adherence BAASIS | 12 months
  To assess the patient-adherence of therapy based on the BAASIS questionnaire
Adherence prescriptions | 12 months
  To assess the patient-adherence of therapy based on the prescription filled by individual patients, based on electronic health-care record.

CONTACTS AND LOCATIONS:
Overall Officials: László Piros, MD, PhD, Principal Investigator — Semmelweis University, Department of Surgery, Transplantation and Gastroenterology, Budapest, Hungary
Locations (2):
- Semmelweis University, Department of Surgery, Transplantation and Gastroenterology, Budapest, Hungary
- University Medical Center Ljubljana, Division of Internal Medicine, Department of Gastroenterology, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No